CLINICAL TRIAL: NCT06176690
Title: Constitutive IL7R (C7R) Modified Banked Allogeneic CD30 Chimeric Antigen Receptor Epstein-Barr Virus-Specific T Lymphocytes (CD30.CAR-EBVSTs) in Patients With Relapsed or Refractory CD30-Positive Lymphomas
Brief Title: Constitutive IL7R (C7R) Modified Banked Allogeneic CD30.CAR EBVSTS for CD30-Positive Lymphomas
Acronym: CABAL2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Premal Lulla, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-56523, CABAL2
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: CD30-Positive Diffuse Large B-Cell Lymphoma; Anaplastic Large Cell Lymphoma, T Cell and Null Cell Type; Anaplastic Large Cell Lymphoma, ALK-Positive; Peripheral T-cell Lymphoma; Anaplastic Large Cell Lymphoma, ALK-negative; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: CD30-Positive Lymphoma; Hodgkin lymphoma; non-Hodgkin lymphoma; CD30 CAR
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Peripheral; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Phase (Experimental): Four dose levels will be evaluated based on safety data from our current study of CD30 CAR T cells.
  Cohorts of three patients will be enrolled at each dose level The dose is based on the number of CD.30 CAR-EBVT-expressing cells administered.
  The total number of dose levels evaluated will depend upon toxicities experienced. Dose level cohorts will be numbered sequentially.
  * Dose Level 1: 4 × 10^7 C7R.CD30.CAR-EBVST cells
  * Dose Level 2: 1 × 10^8 C7R.CD30.CAR-EBVST cells
  * Dose Level 3: 4 × 10^8 C7R.CD30.CAR-EBVST cells
  * Dose Level 4: 8 × 10^8 C7R.CD30.CAR-EBVST cells
  Interventions: Biological: C7R.CD30.CAR-EBVST cells

INTERVENTIONS:
Biological: C7R.CD30.CAR-EBVST cells — The dose is based on the number of CD30.CAR- expressing cells. In our previous study the highest dose was 4 × 10^8 cells/m2 and we did not reach an MTD. On Day 0, patients will receive their planned dose of investigational T cell product by IV infusion over approximately 1 to 10 minutes in an expected volume of 1 to 50 mL.
  Other Names: Allogeneic CR7.CD30 Chimeric Antigen Receptor Epstein-Barr Virus-Specific T Lymphocytes

SUMMARY:
This study involves patients that have a cancer called diffuse large B cell lymphoma (DLBCL), Natural killer/T-cell lymphoma (NKTL), or classical Hodgkin lymphoma (cHL) (referred to collectively as lymphoma). Patients' lymphoma has come back or not gone away after treatment.

A previous research study at Baylor combined two ways of fighting disease: antibodies and T cells. Antibodies are proteins that bind to bacteria, viruses and other foreign substances to prevent disease. T-cells are special infection-fighting white blood cells that can kill tumor cells or cells infected with bacteria and viruses. Both have shown promise treating cancer, but neither has been strong enough to cure most patients. In the previous study, an antibody called anti-CD30 which is found on the surface of some T-cells and cancer cells, and had been used to treat lymphoma with limited success, was joined to the T-cells through a process called gene transfer, resulting in CD30.CAR T cells.

Another study saw encouraging responses using CD30.CAR T cells made in a lab from a patients' own blood then injected back into the same patient to treat their lymphoma. These cells are termed 'autologous' because they're given back to the original patient.

In an ongoing study, patients were treated with allogeneic CD30.CAR T cells, which are made from healthy donors instead of the patients. The use of allogenic cells avoids a lengthy manufacture time since the products are stored as a bank and available on demand. This ongoing trial has preliminarily shown promising clinical activity with no safety concerns.

With the current study, investigators plan to extend the anti-cancer effects of the CD30.CAR T cell by attaching another molecule called C7R, which has made CAR T cells have deeper and longer anticancer effects in the laboratory. The aim is to study the safety and effectiveness of allogeneic banked CD30.CAR-EBVST cells that also carry the C7R molecule, to learn the side effects of C7R modified CD30.CAR-EBVST cells in lymphoma patients, and to see whether this therapy may help them. As an extra safety step, the C7R containing T cells will also have a marker called iC9. If a patient experiences intolerable side effects from the C7R T cells, they could receive a medication called 'rimiducid' that can eliminate the C7R containing T cells by binding iC9, thereby potentially resolving the side effects. While not yet FDA approved, rimiducid has been tested in patients before without bad side effects.

DETAILED DESCRIPTION:
This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose (1 of 4 different levels) of C7R.CD30.CAR-EBVST cells. Once the lower dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 4 dose levels are studied. If the side effects are too severe, the dose will be lowered or the T cell infusion will be stopped. Both the risks and benefits of this study may be dose related. The investigators don't know the best dose that will provide benefit while minimizing the risks.

To enroll on this study, patients will need to have recovered from toxic effects of previous chemotherapy and not be receiving any other investigational agents. Patients cannot have received an investigational cell therapy or vaccine within the past 6 weeks. Patients cannot have received an investigational small molecule drug within the past 2 weeks.

If patients agree to take part in this study, the investigators will ask the patients to adhere to the following study visits and procedure. After patients have signed the consent form, patients are required to come to the hospital for a series of standard medical screening tests, lymphodepletion chemotherapy, infusion with CD30.CAR-EBVST cell treatment and follow-up visits (See details below).

1. Screening tests Screening tests include:

   * Blood tests [Human Leukocyte Antigen (HLA) testing] to help us identify the best match for patients from the banked CD30.CAR- EBVST cells.
   * Blood tests for viruses such as human immunodeficiency virus [HIV], human T cell lymphotropic virus [HTLV], hepatitis B virus and hepatitis C virus.
   * Tumor biopsy test to check the status of CD30.

   Once the investigators find that patients are eligible for this study, patients will be called for additional screening tests before treatment day. The screening tests include:
   * Physical examination
   * Vital signs tests to measure temperature, pulse, respiratory rate and blood pressure
   * Blood tests to measure blood cells, kidney and liver functions
   * Urine test
   * Pregnancy test for women of child-bearing potential
   * Measurements of tumor by routine imaging studies
2. Lymphodepletion chemotherapy Several studies suggest that the infused T cells need room to be able to multiply and grow to accomplish their functions and that this may not happen if there are too many other T cells in the blood stream. Because of that, if patients have NOT had a bone marrow or stem cell transplant recently, patients will receive treatment with cyclophosphamide and fludarabine (chemotherapy drugs) before patients receive the C7R.CD30.CAR-EBVST cells if patient's doctor thinks this is appropriate. This is called "lymphodepletion". These drugs will decrease the numbers of patients own T cells before the investigators inject the C7R.CD30.CAR-EBVST cells. Although the investigators do not expect any effect on the patients tumor with the dose that the patients will receive, these drugs are part of many regimens that are used to treat lymphoma.
3. Treatment with C7R.CD30.CAR-EBVST cells

   Each patient will receive a total dose of CAR modified T cells as detailed below. Dose level cohorts will be numbered sequentially:
   * Dose Level 1: 4 × 10^7 C7R.CD30.CAR-EBVST cells
   * Dose Level 2: 1 × 10^8 C7R.CD30.CAR-EBVST cells
   * Dose Level 3: 4 × 10^8 C7R.CD30.CAR-EBVST cells
   * Dose Level 4: 8 × 10^8 C7R.CD30.CAR-EBVST cells

   The C7R.CD30.CAR-EBVST cells will be infused via an IV line at the indicated dose. Before patients receive the infusion, they may be given a dose of acetaminophen or anti-histamine (Benadryl for example) to minimize any possible allergic reaction. The investigators will follow patients in the clinic after each infusion for at least 3 hours. The patient will need to stay less than 2 hours away from the Medical Center for 4 weeks after the C7R.CD30.CAR-EBVST cell infusion so the investigator can monitor them for side effects.
4. Follow-up visits:

On follow-up visits after treatment, patients will also receive a series of standard medical tests:

* Physical examination
* Vital sign tests to measure temperature, pulse, respiratory rate and blood pressure
* Blood tests to measure blood cells, kidney and liver functions
* Urine tests (if clinically necessary)
* Pregnancy test for women of child-bearing potential (if clinically necessary)
* Measurements of tumor by routine imaging studies

After infusion of C7R.CD30.CAR-EBVST cells, the patients blood will be collected on follow-up visits at week 1, week 2, week 3, week 4, week 8, every 3 months for 1 year, every 6 months for 4 more years then yearly for a total of 15 years (all of these dates are counted from the first infusion). In the event of repeat infusions, for each repeat infusion the calendar will reset, and the follow-up visits will be timed by counting from the date of the most recent T-cell infusion. A tumor biopsy may be done within 4 weeks after the initial C7R.CD30.CAR-EBVST cell infusion. The investigators will also look at any scans or biopsies patients have had as standard of care.

Participants may ask their treating team for a list of potential research costs patients are responsible for and where they are done.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis and clinical course falling into one of the following categories:

   1. Hodgkin lymphoma
   2. CD30+ aggressive B-cell lymphoma
   3. ALK-negative anaplastic T cell lymphoma or other peripheral T- cell lymphoma
   4. ALK-positive anaplastic T cell lymphoma
2. CD30-positive tumor as assayed in a CLIA certified Pathology Laboratory.
3. Age 12 to 75.
4. Bilirubin less than or equal to 2 times the upper limit of normal (except for Gilbert syndrome, where the criteria will be Bilirubin less than or equal to 3 times the upper limit of normal).
5. AST less than 3 times the upper limit of normal.
6. Estimated GFR > 70 mL/min.
7. Pulse oximetry of > 90% on room air
8. Karnofsky or Lansky score of > 60%.
9. Recovered from all acute non-hematologic toxic effects of all prior chemotherapy.
10. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.
11. Informed consent explained to, understood by and signed by patient or guardian. Patient or guardian given a copy of the informed consent form.

Exclusion Criteria:

1. Received an investigational cell therapy or vaccine within the past 6 weeks.
2. Received an investigational small molecule drug within the past 2 weeks.
3. Received CD30 antibody-based therapy within the previous 4 weeks.
4. History of hypersensitivity reactions to murine protein-containing products.
5. Pregnant or lactating.
6. Tumor in a location where enlargement could cause airway obstruction (determined at the investigators' discretion).
7. Current use of systemic corticosteroids at a dose equivalent to or higher than 10 mg/day of prednisone.
8. Active significant, uncontrolled bacterial, viral or fungal infection.
9. Symptomatic cardiac disease (NYHA Class III or IV disease).

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-07-27 (Estimated); Study Completion 2043-06-27 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity rate (DLT) by CTCAE 5.0 | 28 days
  Any Grade 5 event, / Non-hematologic dose-limiting toxicity is any Grade 3 or Grade 4 non-hematologic toxicity that fails to return to Grade 2 within 72 hours, / Grade 2-4 allergic reaction to T-Cells, / Grade 3-4 GVHD, /Hematologic dose limiting toxicity is defined as any Grade 4 hematologic toxicity that fails to return to Grade 2 or baseline (whichever is more severe) within 14 days or within 28 days for patients with evidence of bone marrow disease.

SECONDARY OUTCOMES:
Rate of Anti-Tumor effect Objective Response (OR) | 6 to 8 weeks post CTL infusion
  Objective response rate is defined as complete response and partial response
Duration of response | Up to 5 years
  Response duration will be measured from the time of initial response until documented tumor progression.
Stable disease (SD) rate | 6 to 8 weeks post CTL infusion
  SD will be defined as the proportion of patients that have stable disease
Duration of SD | Up to 5 years
  Stable disease is measured from the start of the treatment until the criteria for progression are met.
Progression free survival (PFS) | Up to 5 years
  PFS is defined as the time from treatment until objective tumor progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Lulla, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas